CLINICAL TRIAL: NCT00858429
Title: Dose Escalating Study of Yttrium 90 Microspheres (TheraSphere) With Capecitabine (Xeloda) for Intrahepatic Cholangiocarcinoma or Metastatic Disease to the Liver
Brief Title: Yttrium Y 90 Glass Microspheres and Capecitabine in Treating Patients With Liver Cholangiocarcinoma or Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mary Mulcahy, Principal Investigator, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 08I5; NU-08I5; STU00007062; NCI-2009-01122 (Other: NCI CTRP#)
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2018-01

CONDITIONS: Liver Cancer; Metastatic Cancer
Keywords: advanced adult primary liver cancer; liver metastases; adult primary cholangiocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; doxifluridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (capecitabine, Y90) (Experimental): 2,000mg/m2 capecitabine +110 Y90
  Interventions: Drug: capecitabine; Radiation: yttrium Y 90 glass microspheres
- Cohort 2 (capecitabine , Y90) (Experimental): 2,000mg/m2 capecitabine + 130 Y90
  Interventions: Drug: capecitabine; Radiation: yttrium Y 90 glass microspheres
- Cohort 3 (capecitabine, Y90) (Experimental): 2,000mg/m2 Capecitabine + 150 Y90
  Interventions: Drug: capecitabine; Radiation: yttrium Y 90 glass microspheres
- Cohort 4 (capecitabine, Y90) (Experimental): 2,000 mg/m2 capecitabine = 170 Y90
  Interventions: Drug: capecitabine; Radiation: yttrium Y 90 glass microspheres

INTERVENTIONS:
Drug: capecitabine — 1000 mg/m2 twice daily, for 14 consecutive days followed by a 7 day treatment free rest period for cycles 1, 2 and 3.
  Other Names: C14H15FN3O7; prodrug of 5'-deoxy-5-fluorouridine (5'-DFUR)
Radiation: yttrium Y 90 glass microspheres — The amount of radioactivity required to deliver the desired dose to the liver is calculated using a formula. The dose depends on the cohort upon which the patient is enrolled. Y90 is administered during Cycle #2 on days 1-7.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. Specialized radiation therapy, such as yttrium Y 90 glass microspheres that deliver a high dose of radiation directly to the tumor, may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Capecitabine may also make tumor cells more sensitive to radiation therapy.

PURPOSE: This phase I trial is studying the side effects and best dose of yttrium Y 90 glass microspheres when given together with capecitabine in treating patients with liver cholangiocarcinoma or liver metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Establish the maximally tolerated dose of yttrium Y 90 glass microspheres in combination with capecitabine in patients with intrahepatic cholangiocarcinoma or liver metastases.
* Characterize the toxicity of this regimen in these patients.
* Determine the time to tumor progression in these patients.

OUTLINE: This is a dose escalation study of yttrium Y 90.

Patients receive oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients also receive yttrium Y 90 glass microspheres by intra-arterial hepatic infusion on days 1-7 of course 2.

After completion of study therapy, patients are followed every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Intrahepatic cholangiocarcinoma
  * Metastatic cancer confined to the liver
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension as ≥ 20 mm by conventional techniques or as ≥ 10 mm by spiral CT scan
* Must have tumor volume ≤ 50% of total liver volume based on visual estimation

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* Serum creatinine ≤ 2.0 mg/dL
* Serum bilirubin ≤ 1.5 times upper limit of normal
* Albumin ≥ 2.0 g/dL
* No baseline symptoms or laboratory values > grade 2 in severity by NCI CTCAE v 3.0 criteria
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No malabsorption syndrome
* No severe liver dysfunction or pulmonary insufficiency
* No complete occlusion of the main portal vein
* No contraindication to iodine-based contrast agents
* No contraindication to hepatic artery catheterization (e.g., vascular abnormalities or bleeding diathesis)
* No prior unanticipated severe reaction to fluoropyrimidine therapy, known hypersensitivity to fluorouracil, or known dihydropyrimidine dehydrogenase deficiency

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the liver
* No more than 2 prior therapies for metastatic disease to the liver
* No prior intervention to or compromise of the Ampulla of Vater
* At least 4 weeks since prior and no concurrent sorivudine or brivudine
* No concurrent cimetidine

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2014-03-19 (Actual); Study Completion 2014-07-08 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose of yttrium Y 90 | During treatment and any time up to 6 weeks post-treatment
Toxicity profile of yttrium Y 90 | During treatment and up to 30 days post-treatment
  Toxicity will be defined as number of adverse events related to treatment experienced during treatment
Time to tumor progression | At time of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Mary Mulcahy, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Northwestern University, Chicago, Illinois, United States